CLINICAL TRIAL: NCT05893810
Title: Bacterial Decolonization to Prevent Radiation-induced Oral Mucositis: A Randomized Controlled Trial and Quality of Life Assessment
Brief Title: Bacterial Decolonization to Prevent Radiation-induced Oral Mucositis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NPC-RIMO
Record Dates: First submitted 2023-05-23; First posted 2023-06-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-05

CONDITIONS: Nasopharyngeal Carcinoma; Radiation-induced Oral Mucositis; Bacterial Colonization; Quality of Life
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): The purpose of this study is to determine whether bacterial decolonization of the nares prior to treatment with radiotherapy (RT) for patients with nasopharyngeal carcinoma, can prevent radiation-induced oral mucositis(RIOM) and improve quality of life.
  Interventions: Drug: Mupirocin Ointment
- Control (No Intervention): Patients in the control arm will be treated according to standard of care.

INTERVENTIONS:
Drug: Mupirocin Ointment — Patients in the intervention arm will receive a decolonization regimen, consisting of intranasal mupirocin ointment to be applied twice daily to the nares
  Arms: Treatment Arm

SUMMARY:
The purpose of this study is to determine whether bacterial decolonization of the nares prior to treatment with radiotherapy (RT) for patients with nasopharyngeal carcinoma, can prevent high-grade radiation-induced oral mucositis (RIOM) and improve quality of life.

This study is being conducted because a randomized clinical trials form Yana Kost et al. have found bacterial decolonization in the nose prior to initiation of RT was effective for prevention of acute radiation dermatitis.

Patients in the treatment arm will receive pretreatment with mupirocin ointment to the nares while patients in the control arm will receive standard of care treatment. Bacterial cultures will be taken from the nares and mouth, and participants will also complete a quality of life questionnaire before and after RT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed nasopharyngeal carcinoma
2. No evidence of distant metastasis (M0)
3. ECOG (Eastern Cooperative OncologyGroup) scale 0-1
4. 18-70 years old

Exclusion Criteria:

1. Previous or existing mental or cognitive impairment;
2. Patients with other malignant tumors at the same time;
3. Have received bacterial decolonization therapy;
4. Oral mucositis or ulcers existed before radiotherapy.
5. Prior RT to the region of interest

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
High-grade radiation-induced oral mucositis | radiation-induced oral mucositis(graded by the RTOG) will be assessed at the last treatment session (study week depends on patient's length of treatment, but ranges from 6 weeks to 8 weeks)
  Grade 3 or higher radiation-induced oral mucositis according to RTOG

SECONDARY OUTCOMES:
High-grade radiation dermatitis | Radiation dermatitis (graded by the CTCAE) will be assessed at the last treatment session (study week depends on patient's length of treatment, but ranges from 6 weeks to 8 weeks)
  Grade 3 or higher radiation-induced dermatitis according to RTOG
Quality of Life according QLQ-H&N43 | Quality of Life (according QLQ-H&N43) will be assessed at the last treatment session (study week depends on patient's length of treatment, but ranges from 6 weeks to 8 weeks)
  EORTC QLQ-H&N43

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kost Y, Deutsch A, Mieczkowska K, Nazarian R, Muskat A, Hosgood HD, Lin J, Daily JP, Ohri N, Kabarriti R, Shinoda K, McLellan BN. Bacterial Decolonization for Prevention of Radiation Dermatitis: A Randomized Clinical Trial. JAMA Oncol. 2023 Jul 1;9(7):940-945. doi: 10.1001/jamaoncol.2023.0444. PMID 37140904
- [Derived] Liao Z, Xiong X, Zhao L, Zhang Z, Guan C, Zhang L, Zhong F, Rao J, Wang X, Xiao Y, Gong X, Huang SH, Li J, Lu T. Bacterial Decolonization With Mupirocin Ointment for Acute Radiation Oral Mucositis Prevention: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2025 Oct 1;11(10):1141-1149. doi: 10.1001/jamaoncol.2025.2361. PMID 40773220